CLINICAL TRIAL: NCT04436770
Title: Medical Recovery and Social Reintegration for Post-stroke Patients With Sequelae Using Virtual Reality
Brief Title: Medical Recovery and Social Reintegration for Post-stroke Patients Using Virtual Reality
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic
Sponsor: Transilvania University of Brasov (Other)
Collaborators: Spitalul Clinic de Psihiatrie si Neurologie Brasov (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 13/8.02.2018
Record Dates: First submitted 2020-06-11; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Stroke Sequelae
Keywords: Virtual Reality; Physiotherapy; Recovery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Standard physiotherapy and OT
  Interventions: Other: Standard Physiotherapy
- Experimental (Experimental): Virtual Reality Therapy and OT
  Interventions: Other: Non-immersive virtual reality therapy

INTERVENTIONS:
Other: Non-immersive virtual reality therapy — Non-immersive Virtual Reality (VR) therapy exercises, based on assessment, and occupational therapy exercises, for upper extremity or lower extremity.
  For the upper extremity, daily, from 20-40 to minutes of VR therapy plus 20-40 minutes of occupational therapy exercises, according to the patient's capacity of VR training, as entire therapy for upper extremity don't exceed 60 minutes.
  For the lower extremity, from 20-40 to minutes of VR therapy plus 20-40 minutes of occupational therapy exercises, according to the patient's capacity of VR training, as entire therapy for the lower extremity don't exceed 60 minutes.
  The protocol for occupational therapy exercises for the hand included the use of the Canadian plate, thick and thin grip training, lateral and palmar pinch as well as wrist extensor strengthening tasks.
  For the ankle and foot, analytical and dexterity exercises using Mirror therapy and alone were used.
  Other Names: Occupational therapy exercises
  Arms: Experimental
Other: Standard Physiotherapy — Standard physiotherapy program, based on assessment, plus occupational therapy exercises, for upper extremity or lower extremity.
  For the upper extremity, daily, 30 minutes of standard physiotherapy plus 30 minutes of occupational therapy exercises.
  For the lower extremity, daily, 30 minutes of standard physiotherapy plus 30 minutes of occupational therapy exercises.
  The protocol for occupational therapy exercises for the hand included the use of the Canadian plate, thick and thin grip training, lateral and palmar pinch as well as wrist extensor strengthening tasks.
  For the ankle and foot, analytical and dexterity exercises were used.
  Other Names: Occupational therapy exercises
  Arms: Control Group

SUMMARY:
Application of Virtual Reality therapy and occupational therapy versus and standard physiotherapy and occupational therapy to patients with post-stroke sequelae, using specifical assessment tools, standard physiotherapy and occupational therapy programs.

DETAILED DESCRIPTION:
1. Initial and final clinical and functional evaluation of patients with post-stroke sequelae, storage and use of data obtained.
2. Collection and access of demographic and clinical data of patients included in the study (respecting the principle of confidentiality and non-publication of personal data) only by staff involved in the research project and working in the Clinical Hospital of Psychiatry and Neurology in Brasov.
3. Application of Virtual Reality therapy and occupational therapy versus and standard physiotherapy and occupational therapy to patients who meet the criteria for inclusion in the study (scapulohumeral flexion and abduction of at least 20 degrees, elbow flexion of at least 20 degrees, hip and knee flexion of at least 20 degrees, without severe aphasia or severe behavioural/cognitive disorders).
4. Use of data obtained from the application of Virtual Reality therapy at home, through Telerehabilitation, if patients procure alone or through sponsorship/donation the equipment necessary to continue the Virtual Reality therapy program at home, taking into account that the technology purchased through the project allows this.

ELIGIBILITY:
Inclusion Criteria:

1. stroke survivors after the acute phase, at least 6 weeks post-stroke;
2. stroke survivors within no more than 4 years after stroke,
3. at least 30-degree flexion and scapulohumeral abduction against gravity.
4. elbow flexion of at least 30 degrees
5. hip flexion of at least 30 degrees
6. knee flexion of at least 30 degrees

Exclusion Criteria:

1. no severe cognitive impairments,
2. no global or transcortical sensory aphasia,
3. no other dysfunctions in the upper extremity such as surgery, fractures, shoulder arthritis or severe pain,
4. no other dysfunctions in the lower extremity such as surgery, fractures, arthritis or severe pain,
5. without anaemia
6. without atrial fibrillation
7. without NYHA class IV heart failure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of patients for whom tailored Virtual Reality therapy is more efficient than standard tailored physiotherapy in the recovery of post-stroke sequelae. | One year since the beginning of the research
  Determining the factors and parameters that influence or enhance post-stroke recovery capacity using new recovery methods, such as non-immersive virtual reality.
  The assessment tools are: the Fugl-Meyer assessment for the upper extremity (FMUE), Fugl-Meyer assessment for the lower extremity (FMLE), the Modified Rankin Scale (MRS), the Functional Independence Measure (FIM), the Active Range of Motion (AROM), the Manual Muscle Testing (MMT), the Modified Ashworth Scale (MAS), the Functional Reach Test (FRT), and Timed Up and Go Test (TUG).
  The patients are assessed by recovery medical doctors (physiatrists) regarding FIM, MAS and MRS. While FMUE, FMLE, AROM, MMT, FRT, TUG are assessed by trained physiotherapists, with at least 5 years of experience in stroke sequelae physiotherapy and evaluation.

SECONDARY OUTCOMES:
The number of patients for whom heart disease and other elderly condition, age or gender are influencing the capacity to the recovery of post-stroke patients. | One year since the beginning of the research
  Collecting data related to age, gender, time after stroke, other conditions present (such as hypertension, dyslipidemia, diabetes, ischemic coronary disease, etc.) and determining the links between post-stroke recovery capacity and these factors using statistical software programs and analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital of Psychiatry and Neurology, Brasov, Brașov County, Romania

IPD SHARING:
Plan to Share IPD: No